CLINICAL TRIAL: NCT00928005
Title: Diet and Exercise in Type 2 Diabetes and Prediabetes
Brief Title: Evaluating the Effects of a Diet and Exercise Program in People With Type 2 Diabetes or Prediabetes: (The SHAPE3 Study)
Acronym: SHAPE3
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Kerry Stewart, Professor of Medicine, National Heart, Lung, and Blood Institute (NHLBI)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 666; 1R01HL086026-01A2 (NIH)
Record Dates: First submitted 2009-06-23; First posted 2009-06-25 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-04

CONDITIONS: Overweight; Obesity; Type 2 Diabetes; Prediabetes
Keywords: Weight loss diet; Exercise training; Type 2 diabetes; Prediabetes; Cardiovascular health
MeSH Terms: conditions — Overweight; Obesity; Diabetes Mellitus, Type 2; Prediabetic State | interventions — Diet, Reducing; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Weight loss diet (Active Comparator): Participants will follow a low-calorie, low-fat weight loss diet for 6 months.
  Interventions: Behavioral: Weight loss diet
- Weight loss diet plus exercise (Active Comparator): Participants will follow a low-calorie, low-fat weight loss diet plus participate in a supervised exercise training program for 6 months.
  Interventions: Behavioral: Weight loss diet plus exercise

INTERVENTIONS:
Behavioral: Weight loss diet — The weight loss diet will follow the American Diabetes Association guidelines and be nutritionally balanced with a reduced saturated fat content.
  Arms: Weight loss diet
Behavioral: Weight loss diet plus exercise — The supervised exercise training sessions will take place three times a week for 6 months. Each session will last 1 to 1 ½ hours and will include aerobic exercise and weight training.
  Arms: Weight loss diet plus exercise

SUMMARY:
Type 2 diabetes and prediabetes, which are mainly caused by a lack of physical activity and excess weight, put people at an increased risk of cardiovascular disease. This study will compare the effects of a weight loss diet versus a weight loss diet plus an exercise program on body composition and cardiovascular factors that are early predictors of future cardiovascular disease in overweight and obese people with type 2 diabetes and prediabetes.

DETAILED DESCRIPTION:
Type 2 diabetes and prediabetes are conditions that are largely caused by excess weight and physical inactivity. These conditions have adverse effects on heart and blood vessel structure and function, including left ventricular diastolic dysfunction, endothelial vasodilator dysfunction, and increased vascular stiffness, each of which increase the risk of cardiovascular disease. Reducing the amount of calories consumed and increasing physical activity are both important factors for losing weight, increasing fitness, and improving blood glucose control. However, little research has been conducted on the combined effects of diet and exercise on general and abdominal obesity, fitness, heart and blood vessel structure and function, and heart disease risk factors. The purpose of this study is to determine whether people who follow a diet program plus an exercise program experience better improvements in body composition and cardiovascular health than people who follow only a diet program.

This study will enroll people who are overweight or obese and have type 2 diabetes or prediabetes. Participants will attend a baseline study visit and complete blood pressure measurements; muscle strength measurements; a treadmill test to evaluate cardiovascular fitness; an echocardiogram to obtain images of the heart; tests to measure blood vessel function; a dual energy x-ray absorptiometry (DEXA) scan to measure body fat, muscle tissue, and bone density; questionnaires to assess physical activity levels, quality of life, and mood; and a blood collection. A portion of blood will be stored for future genetic testing. Women will also provide a urine sample for pregnancy testing. Participants will also keep a food diary for 3 days. Participants will then be randomly assigned to either a weight loss diet group or a weight loss diet plus exercise group. All participants will attend study visits with a dietitian for weight loss counseling once a week during Months 1 and 2, and every other week in Months 3 through 6. At each of these visits, participants' weight will be measured. Blood pressure measurements will also occur at least once a month.

Participants who are assigned to the diet plus exercise group will also attend a supervised exercise session three times a week for 6 months. Each session will last 1 to 1 ½ hours and will include aerobic exercise and weight training. Participants who have diabetes or who are receiving medication to control their blood sugar will have their blood sugar measured before and after exercising, based on study staff recommendations. At the end of Month 6, all participants will attend a study visit for repeat baseline testing.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) 25-42kg/m^2
* Type 2 diabetes or prediabetes

Exclusion Criteria:

* Currently smokes
* History or evidence of cardiovascular disease or other major chronic illness
* Currently exercising regularly or following a weight loss diet
* Uncontrolled high blood pressure
* Any illness that would prevent participation in a moderate-intense exercise program
* Pregnant
* Substance abuse
* Use of insulin

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2009-07; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Cardiovascular structure and function | Measured at 6 months

SECONDARY OUTCOMES:
Body composition | Measured at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Kerry J Stewart, EDD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States